CLINICAL TRIAL: NCT00287807
Title: Self-monitoring of Blood Glucose in Patients With Type 2 Diabetes Mellitus Who Are Not Using Insulin. A Randomized Controlled Trial
Brief Title: Effect of Self-monitoring of Blood Glucose in Patients With Type 2 Diabetes Mellitus Not Using Insulin
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medical Research Foundation, The Netherlands (Other)
Collaborators: Langerhans Foundation, the Netherlands (Other)
Responsible Party: Principal Investigator, Nanne Kleefstra, MD PhD, Medical Research Foundation, The Netherlands
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IC-06-02-SL
Record Dates: First submitted 2006-01-30; First posted 2006-02-07 (Estimated); Last update posted 2011-09-26 (Estimated); Status verified 2011-09

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes mellitus, type 2; Blood Glucose Self-Monitoring; life style
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Blood Glucose Self-Monitoring

INTERVENTIONS:
Behavioral: Self-monitoring of blood glucose (SMBG) — 2 times a week (one in weekend and one during week) self measurement of blood glucose: fasting and three times post prandial

SUMMARY:
Self-monitoring of blood glucose (SMBG) is one of the important instruments in diabetes management. Most patients with type 1 diabetes and patients with type 2 using insulin, frequently measure their blood glucose in case of possible hypoglycemia, but also to evaluate the insulin treatment and get information about how to change the insulin regimen, if necessary. Without SMBG it is almost impossible to achieve this goal.

The purpose of this study is to determine if self-monitoring in patients with type 2 diabetes not using insulin results in better glycemic control.

DETAILED DESCRIPTION:
Study Objectives:

Primary: What is the effect of SMBG in patients with type 2 diabetes who are not using insulin on Glycemic control (as measured with glycosylated hemoglobin (HbA1c)?

Secondary: What is the effect of SMBG in patients with type 2 diabetes who are not using insulin on the following parameters:

* Health status
* Diabetes related complaints
* Patient satisfaction
* Cumulative incidence of (necessity to start) insulin therapy / maximum dosage of oral blood glucose lowering drugs
* Dosage of oral blood glucose lowering drugs
* Bodyweight (BMI)

Two treatment protocols are proposed. Treatment A consists of self-monitoring of blood glucose and treatment B consists of usual care. Patients in the A-group are instructed to measure their blood glucose values 4 times a day (1 fasting plasma glucose concentration and 3 post-meal glucose concentrations), two times a week, on one week day, and one weekend day (no more, no less). Patients should record these glucose values in a diary. Patient will get one page with information in Dutch. No further education than for handling the device and interpreting the values is given, so that besides this intervention, there will be no differences compared with the control group like other forms of education.

The duration fo the trial will be 12 months.

ELIGIBILITY:
Inclusion criteria:

* Type 2 diabetes
* HbA1c 7 - 8,5% at previous and present annual check-up
* Use of 1 or 2 different oral blood glucose lowering drugs
* In case of two oral blood glucose lowering drugs, they should not both have a maximum dosage
* Sufficient knowledge of the Dutch language to understand the requirements for the study

Exclusion criteria:

* Change in oral blood glucose lowering drugs in the past three months
* Use of insulin
* Use of device for self-monitoring of blood glucose at the start of the study, or in the preceding 6 months

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2006-02; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Glycemic control; HbA1c at baseline, 3 months, 6 months, 9 months and 1 year (endpoint) | baseline, 3 months, 6 months, 9 months and 1 year (endpoint)

SECONDARY OUTCOMES:
Quality of life; score on scale at baseline, 6 months and endpoint | baseline, 6 months and endpoint
Diabetes related complaints; score at baseline, 6 months and endpoint | baseline, 6 months and endpoint
Treatment satisfaction; score on scale at baseline, 6 months and endpoint | baseline, 6 months and endpoint
Incidence of (necessity to start) insulin therapy; at endpoint | anywhere during the study
dosage of oral blood glucose lowering drugs; at baseline, 6 months and endpoint | baseline, 6 months and endpoint
bodyweight; Bodymass index at baseline and endpoint | baseline and endpoint

CONTACTS AND LOCATIONS:
Overall Officials: Henk J Bilo, MD; PhD, Principal Investigator — Isala Clinics, medical research foundation
Locations (1):
- Isala Clinics, Zwolle, Netherlands